CLINICAL TRIAL: NCT01753180
Title: A 2-stage Study to Evaluate Single Doses of MZ-004 at Different Dose Levels in Patients With Chronic Total Occlusions. Stage 1: Open Label Training Stage. Stage 2: Double-blind, Randomized, Placebo-Controlled Stage
Brief Title: Total Occlusion Study in Coronary Arteries - 5
Acronym: TOSCA-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matrizyme Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTO-201
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Coronary Total Occlusions
Keywords: CTO; PCI; Angioplasty
MeSH Terms: interventions — Collagenases; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- collagenase (Experimental)
  Interventions: Biological: collagenase
- saline (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Biological: collagenase — Local intra-coronary administration of MZ-004 at or into the CTO
  Other Names: MZ-004
  Arms: collagenase
Drug: saline — Local intra-coronary administration of saline at or into the CTO
  Arms: saline

SUMMARY:
A prospective, multi-center, double blind, 2 stage, placebo-controlled, phase II study, evaluating acute intra-coronary injected collagenase prior to routine standard-of-care percutaneous revascularization procedures in subjects with chronic total coronary artery occlusions (CTOs).

ELIGIBILITY:
Inclusion Criteria:

* Male or females patients > 18 years of age who has a clinically driven, planned PCI of the target CTO, in a major epicardial coronary artery, without planned revascularization of other coronary stenosis/stenoses in major epicardial segments.
* Target CTO must be greater than or equal to 3 calendar months prior to Screening
* Target CTO must meet protocol defined criteria for entry
* Patient is receiving a course of optimal anti-ischemic medical therapy (at least 2 anti-anginal agents or the maximum tolerated anti-anginal therapy)

Exclusion Criteria:

* Documented chest radiation exposure > 4.0 Gray within 8 weeks of Day 0
* Target vessel is not an occluded stent, saphenous vein graft
* Patient had ACS < 4 weeks from Screening, attributable to any coronary vessel
* Patient has non-healed dissection plane extending to a point adjacent to the coronary lumen distal to the target CTO
* Patient has a known or suspected target vessel perforation within 30 days of Day 0
* Angiographic exclusion criteria as defined in the protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Anterograde PCI success rate for patients with a target CTO | Day 1 of study procedures
  To assess the PCI success rates in CTOs that have failed a previous PCI attempt between different doses of MZ-004 and placebo

SECONDARY OUTCOMES:
Total fluoroscopy time | Day 0 and Day 1 of study procedures
  To assess the total fluoroscopy time between patients treated with two different doses of MZ-004 and/or placebo
Total PCI procedural time | Day 1 of study procedures
  To assess the total procedural time between patients treated with two different doses of MZ-004 and/or placebo
Soft wire crossing | Day 1 study procedures
  To assess the percentage of lesions that are crossed with soft guide wires post study drug administration
Safety | Day 0, Day 1 and Day 2 of study procedures
  To assess the overall safety of the procedure in evaluating treatment emergent adverse events, major adverse cardiac events, radiation exposure, angiographic complications, ECGs, vital signs and clinical laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Buller, Dr., Principal Investigator — St. Michael's Hospital, Toronto, Ontario, Canada
Locations (13):
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CHUM Hotel Dieu, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre de recherche de l'Institut Universitaire de Pulmonologie et Cardiologie de Quebec, Ste. Foy, Quebec
- Shaare Zedek Medical Center, Jerusalem, Israel
- Academic Medical Center, Amsterdam, Netherlands